CLINICAL TRIAL: NCT05203263
Title: Evaluation of the Tolerance and the Mode of Administration of Cyto-selective Difluoroethane-based Cryotherapy in the Treatment of Brown Spots
Brief Title: Tolerance and Mode of Administration of Cyto-selective Cryotherapy Treatments in Face Brown Spots: Proof of Concept
Acronym: AGILE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cryonove Pharma (Industry)
Collaborators: Dermatech (Industry); CEISO (Industry); INNOVSOLUTION (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: (CS4_2) AGILE 2 N° 21D588A0002
Record Dates: First submitted 2021-12-13; First posted 2022-01-24 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-01

CONDITIONS: Solar Lentigo
Keywords: Lentigo; Melanosis; melanocyte; melanosome; Hyperpigmentation; Pigmentation Disorders; Skin Diseases
MeSH Terms: conditions — Lentigo; Melanosis; Hyperpigmentation; Pigmentation Disorders; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Condition 1 : Prototype (810A-v1) and Frequency of application 1 (Experimental): Application of the prototype (810A-v1) at Day 0, Day 1, Day 2, Day 3, Day 4 and Day 5.
  Interventions: Device: (810A-v1) device prototype
- Condition 2 :Prototype (810B-v1) and Frequency of application 1 (Experimental): Application of the prototype (810B-v1) at Day 0, Day 1, Day 2, Day 3, Day 4 and Day 5.
  Interventions: Device: (810B-v1) device prototype
- Condition 3 : Prototype (810A-v1) and Frequency of application 2 (Experimental): Application of the prototype (810A-v1) at Day 0, Day 7, Day 14, Day 21, Day 28 and Day 35.
  Interventions: Device: (810A-v1) device prototype
- Condition 4 : Prototype (810C-v1) and Frequency of application 2 (Experimental): Application of the prototype (810C-v1) at Day 0, Day 7, Day 14, Day 21, Day 28 and Day 35.
  Interventions: Device: (810C-v1) device prototype
- Condition 5 : Prototype (810C-v1) and Frequency of application 3 (Active Comparator): Application of the prototype (810C-v1) at Day 0, Day 14, Day 28, Day 42, Day 56 and Day 70.
  Interventions: Device: (810C-v1) device prototype

INTERVENTIONS:
Device: (810A-v1) device prototype — Sequence with Serial Number from (810-v1 101) to (810-v1 140). Application on brown spots located on the face (6 treatments during the study).
  Arms: Condition 1 : Prototype (810A-v1) and Frequency of application 1; Condition 3 : Prototype (810A-v1) and Frequency of application 2
Device: (810B-v1) device prototype — Sequence with Serial Number (810-v1 141) to (810-v1 160). Application on brown spots located on the face (6 treatments during the study).
  Arms: Condition 2 :Prototype (810B-v1) and Frequency of application 1
Device: (810C-v1) device prototype — Sequence with Serial Number (810-v1 161) to (810-v1 200). Application on brown spots located on the face (6 treatments during the study).
  Arms: Condition 4 : Prototype (810C-v1) and Frequency of application 2; Condition 5 : Prototype (810C-v1) and Frequency of application 3

SUMMARY:
Solar lentigos or lentigines are harmless patch of darkened skin, of different sizes and colors, due to the exposure to UV radiation. They are very common, especially in people over the age of 40 years old. Solar lentigines appears as clusters of similar lesions on sun-exposed sites, such as the face or the back of the hands.

Conventional cryotherapy is increasingly used to improve the skin appearance and especially to treat lentigo spots. However, the application of conventional cryotherapy is followed by temporary side effects including pain at application, hypo- and hyperpigmentation, crust, scars, burns, erythema... for a few days after administration and that can persist during several months.

In this context, the sponsor has developed a treatment using cyto-selective cryotherapy, that treats only the melanocytes responsable of brown spots while preserving other cells of the epidermis. Several sequences of pulverization of cryogenic gas have been designed. It seems interesting for the sponsor to study some ways of applications of the selected sequences. i.e. 5 conditions evaluated) that could be used for the treatment of lentigos with the same clinical benefit and with better safety results for patients .

(CS4_2) proof of concept, interventional, monocentric, randomized and double blinded study, aims to evaluate the tolerance and the mode of administration of cyto-selective difluoroethane-based cryotherapy in the treatment of brown spots.

The main objective of the study is to evaluate the tolerance and to adjust the mode of administration of 3 different cryotherapy treatments (3 prototypes) applied on the brown spots of the face. Each treatment corresponds to a specific sequence of a cryogenic spray.

DETAILED DESCRIPTION:
Prototypes (810A-v1), (810B-v1) and (810C-v1) will be applied on brown spots located on the face. Regarding the randomization list, each spot will be treated by a defined prototype / device (same prototype /device will be used to treat the same spot all along the study).

Each spot will be treated 6 times during the study:

* At Day 0, Day 1, Day 2, Day 3 Day 4 and Day 5 for the prototypes (810A-v1) (condition 1) and (810B-v1) (condition 2).
* At Day 0, Day 7, Day 14, Day 21, Day 28 and Day 35 for the prototypes (810A-v1) (condition 3) and (810C-v1) (condition 4).
* At Day 0, Day 14, Day 28, Day 42, Day 56 and Day 70 for the prototype (810C-v1) (condition 5, considered as reference).

Prior to any study device application, the dermatologist will assess the adverse events and decide whether the period between two consecutive applications should be extended or not. The dermatologist will verify that the skin has not been treated with cosmetic products (no cream, peeling, dermabrasion, laser treatment... that could interfere with the treatment) and that is dry.

The procedure will take place at the investigation site. An operator previously trained by the dermatologist will apply the study device to the patient's brown spots.

Subjects will lie down and the device will be administered upside down. During the applications, subjects will wear diving goggles (provided by the CRO) to protect the eyes from the cryogenic gas.

Treatments will be stopped when a total of 6 applications for the prototypes will be delivered or as soon as a spot will be considered disappeared by the investigator. Otherwise the study will continue (tolerance report, etc.) until all conditions are completed.

ELIGIBILITY:
Inclusion Criteria:

* Phototype II et III (according with Fitzpatrick scale)
* Featuring brown spots (solar lentigos) on the face ≥ 3mm to 6 mm in diameter (at least 2-3 spots per subject).
* Agreeing not to be exposed to the sun (or artificial UV) during the study.
* Informed, having undergone a general clinical examination attesting to his/her ability to participate in the study.
* Having given written consent for participation in the study.
* No suspicion of carcinoma after investigation by a dermatologist.

Exclusion Criteria:

* Having performed cosmetic treatments (exfoliants, scrubs or self-tanners, facials, UV...) in the month before the start of the study, at the level of the face.
* Having applied a depraving product in the month prior to the start of the study, at the level of the face.
* Having performed cosmetic treatments in a dermatologist (laser, intense pulsed light, peeling, creams, cryotherapy ...), at the level of the face in the last 6 months.
* With dermatosis, autoimmune disease, systemic, chronic or acute disease, or any other pathology that may interfere with treatment or influence the results of the study (people with diabetes or circulatory problems, allergic to cold, Raynaud's syndrome...).
* Receiving treatment by general or local (dermo corticoids, corticosteroids, diuretics ...) likely to interfere with the evaluation of the parameter studied.
* Participating in another study or being excluded from a previous study.
* Unable to follow the requirements of the protocol.
* Vulnerable: whose ability or freedom to give or refuse consent is limited.
* Major protected by law (under guardianship, under curatorship, safeguarding justice...).
* People unable to read and write Ukrainian language.
* Unable to be contacted urgently over the phone.

For female subjects:

* Pregnant woman (or wishing to be pregnant during study) or while breastfeeding.
* A woman, who does not use effective methods of contraception.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline skin hyperpigmentation | - Conditions 1 and 2: Day0, Day1, Day2, Day3, Day4, Day5, Day14 and Day28 - Conditions 3 and 4: Day0, Day1, Day2, Day3, Day7, Day14, Day21, Day28, Day 35 and Day42 - Condition 5 (Ref): Day0, Day1, Day2, Day3, Day14, Day28, Day42, Day56, Day70 and Day84
  This outcome is a tolerance assessment criteria. Clinical evaluation of hyperpigmentation on each selected and treated lentigo spot will be performed by a Dermatologist using the Investigator's Global Assessment likert 6 points scale ranged from 0 to 5: 0=Clear of hyperpigmentation, 1= Almost clear of hyperpigmentation, 2=mild, but noticeable hyperpigmentation, 3=moderate hyperpigmentation (medium brown in quality), 4=severe hyperpigmentation (dark brown in quality), 5= very severe hyperpigmentation (very dark brown, almost black in quality).
Change from baseline skin hypopigmentation | - Conditions 1 and 2: Day0, Day1, Day2, Day3, Day4, Day5, Day14 and Day28 - Conditions 3 and 4: Day0, Day1, Day2, Day3, Day7, Day14, Day21, Day28, Day35 and Day42 -Condition 5 (Ref): Day0, Day1, Day2, Day3, Day14, Day28, Day42, Day56, Day70 and Day84
  This outcome is a tolerance assessment criteria. Clinical evaluation of hypopigmentation on each selected and treated lentigo spot will be performed by a Dermatologist using a likert 5 points scale ranged from 0 to 4: 0=no hypopigmented lesion, 1= very slight area of hypopigmentation of very small size and very slightly fairer than the surrounding skin, 2= slight area of hypopigmentation of small size and slightly fairer than the surrounding skin, 3= moderate : area of hypopigmentation of moderate size and much fairer than the surrounding skin, 4= severe : area of hypopigmentation of large size and much fairer than the surrounding skin.
Change from baseline skin appearance (Edemas, blisters, bubbles, scars, erythema) | - Conditions 1 and 2: Day0, Day1, Day2, Day3, Day4, Day5, Day14 and Day28 - Conditions 3 and 4: Day0, Day1, Day2, Day3, Day7, Day14, Day21, Day28, Day35 and Day42 -Condition 5 (Ref): Day0, Day1, Day2, Day3, Day14, Day28, Day42, Day56, Day70 and Day84
  This outcome is a tolerance assessment criteria. Clinical visual evaluation of selected lentigo spots and surrounded spotless skin area around the spot skin will be performed. A likert scale in 5 points (0 to 4) will be used : 0=none; 1=very mild; 2=mild; 3=moderate; 4=severe.
Change from baseline skin sensation (itching, tingling, burning sensations) | - Conditions 1 and 2: Day0, Day1, Day2, Day3, Day4, Day5, Day14 and Day28 - Conditions 3 and 4: Day0, Day1, Day2, Day3, Day7, Day14, Day21, Day28, Day35 and Day42 -Condition 5 (Ref): Day0, Day1, Day2, Day3, Day14, Day28, Day42, Day56, Day70 and Day84
  This outcome is a tolerance assessment criteria. Clinical visual evaluation of selected lentigo spots and around the spot skin will be performed. A likert scale in 5 points (0 to 4) will be used : 0=none; 1=very mild; 2=mild; 3=moderate; 4=severe.
Post treatment pain | Day 0 (Time1 defined as 15 minutes post-treatment)
  This outcome is a tolerance assessment criteria. The pain of the treatment will be assessed by the VAS (Visual Analogue Scale). Pain intensity is measured in millimeters by the distance from the position of the mark to the "no pain" extremity.
  Based on the distribution of pain VAS (Visual Analogue Scale) scores in postoperative patients, the following bounds were recommended for the assessment of this scale: no pain (0-4mm), mild pain (5-44mm), moderate pain (45-74 mm) and severe pain (75- 100 mm).
Change from baseline skin color | - Conditions 1 and 2: Day0, Day14 and Day28 - Conditions 3 and 4: Day0, Day7, Day14, Day21, Day28, Day35 and Day42 - Condition 5 (Ref): Day0, Day14, Day28, Day42, Day56, Day70 and Day84
  This outcome is a performance assessment criteria. Clinical evaluation of each treated lentigo spot and spotless area (one on face and far from a lentigo spot) will be performed in blinded conditions by a trained assessor by scoring using L'OREAL ColorChart (provided by the Sponsor or L'Oréal) in standardized position and lighting.
Change from baseline spots visibility | - Conditions 1 and 2: Day0, Day1, Day2, Day3, Day4, Day5, Day14 and Day28 - Conditions 3 and 4: Day0, Day1, Day2, Day3, Day7, Day14, Day21, D28, Day35 and Day42 - Condition 5 (Ref): Day0, Day1, Day2, Day3, Day14, Day28, Day42, Day56, Day70 and Day84
  This outcome is a performance assessment criteria. Standardized photographs by C-Cube® acquisition will be taken before the treatment at each visit of each spot using a dermatoscope C-cube (device which allows realizing high resolution skin pictures (10 million pixels 2D capture (UHD)).

SECONDARY OUTCOMES:
Efficacy self-assessment | - Conditions 1 and 2: Day0, Day1, Day2, Day3, Day4, Day5, Day14 and Day28 - Conditions 3 and 4: Day0, Day1, Day2, Day3, Day7, Day14, Day21, Day28, Day35 and Day42 - Condition 5 (Ref): Day0, Day1, Day2, Day3, Day14, Day28, Day42, Day56, Day70 and Day84
  Data will be completed by a questionnaire elaborated by the sponsor and filled in by subjects. It allowed obtaining the subjective appraisal of subject on tested laser act using the following 5-point scale: agree; quite agree; neither agree, nor disagree; quite disagree; disagree.
  The items are the following:
  * The spot seems clearer.
  * The size of the spot seems reduced.
  * The spot seems less visible.

CONTACTS AND LOCATIONS:
Locations (1):
- VIDNOVLENNYA medical center, Zhytomyr, Ukraine